CLINICAL TRIAL: NCT00005780
Title: Pilot Study of Idiotype Vaccine and EPOCH-Rituximab Chemotherapy in Untreated Mantle Cell Lymphoma
Brief Title: Chemotherapy Plus Vaccination to Treat Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Melani, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000133; 00-C-0133; NCT00020215 (obsolete NCT alias)
Record Dates: First submitted 2000-06-03; First posted 2000-06-05 (Estimated); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Mantle Cell Lymphoma; Lymphoma, Mantle Cell
Keywords: Lymphoma Vaccines; Immune Response Against Lymphoma; Molecular Complete Remissions; Novel Treatment Approach; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin; Rituximab; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (Experimental): Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) followed by idiotype vaccine and granulocyte-macrophage colony-stimulating factor (GM-CSF).
  Interventions: Drug: EPOCH-R; Biological: GM-CSF; Biological: Idiotype vaccine

INTERVENTIONS:
Drug: EPOCH-R — EPOCH-R for 6 cycles
  Other Names: Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab
Biological: GM-CSF — Granulocyte-macrophage colony-stimulating factor (GM-CSF) monthly with the vaccine for 5 doses
  Other Names: Sargramostim
Biological: Idiotype vaccine — 1 injection of vaccine monthly for 5 doses

SUMMARY:
This study will evaluate the safety and effectiveness of an experimental cancer vaccine for mantle cell lymphoma a form of cancer of the white blood cells called lymphocytes. Although standard treatments for lymphoma may achieve disease remission, none provides a cure.

Patients with mantle cell lymphoma 18 years and older who have not been treated previously with chemotherapy may participate in this study. Candidates will be screened for eligibility with a medical history and physical examination. Other tests that may be required include blood and urine tests; lung function studies; imaging tests such as magnetic resonance imaging, computed tomography and X-rays; and biopsy (surgical removal of a small tissue sample) of tumor, bone marrow, or other tissue.

Patients enrolled in the study will begin treatment with chemotherapy designed to reduce disease to a minimum that is, to achieve remission or shrink the tumor as much as possible. Chemotherapy will be administered on an outpatient basis over a period of around 12 to 18 weeks in 3-week cycles as follows: prednisone by mouth on days 1 through 5; etoposide, doxorubicin and vincristine intravenously through (a vein) on days 1 through 5; and cyclophosphamide intravenously on day 5. Starting day 6, patients receive no chemotherapy for 16 days. In addition, an antibody called rituximab, which attaches to lymphoma cells and may increase the effectiveness of the chemotherapy, will be given on day 1 of the cycle. Patients will also receive a protein called granulocyte colony-stimulating factor (G-CSF) starting day 6 of the cycle and continuing until the white blood cell count recovers or until day 19. G-CSF is naturally produced by bone marrow and may boost the immune system. The chemotherapy drugs and rituximab are infused through a vein by means of a lightweight portable pump, which patients are taught how to use. Patients are also how taught how to give themselves G-CSF injections under the skin, similar to insulin injections.

The first vaccination will be given at least 3 months after chemotherapy ends and will be repeated every 4 weeks for a maximum of 5 vaccinations. The vaccinations will be given in the clinic. Patients will also receive daily injections of granulocyte-macrophage colony-stimulating factor (GM-CSF), a growth factor naturally produced by bone marrow that can boost the immune system. These injections will be given the day of the vaccination and for the next 3 days.

When vaccine therapy is completed, patients who were treated successfully will be followed with periodic clinic visits for follow-up examinations and tests. Patients in whom the lymphoma did not disappear entirely or who have a recurrence of disease will be advised of further treatment possibilities....

DETAILED DESCRIPTION:
Background:

* Mantle cell lymphoma presents a particular clinical challenge because it is aggressive and incurable with chemotherapy. Thus, novel treatment approaches are needed.
* In follicular center cell lymphomas, another incurable disease, recent evidence suggests that molecular complete remissions may be achieved following idiotype vaccination in patients who have achieved minimal residual disease with combination chemotherapy.
* These results suggest that idiotype vaccines may be able to induce a clinically significant immune response against lymphoma.

Objectives:

* To assess if etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R)/idiotype vaccination is associated with a median progression-free survival consistent with 36 months;
* To assess if rituximab affects generation of T-cell immunity against the idiotype.
* To compare T-cell immunity using two different methods of isolating the idiotype protein.

Eligibility:

* Tissue diagnosis of mantle cell lymphoma.
* Age greater than or equal to 18 years.
* Previously untreated with cytotoxic chemotherapy. All stages of disease.
* Lymph node of greater than or equal to 2 cm accessible for biopsy/harvest or greater than 1000/microl of circulating tumor cells in the blood.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 3.

Design:

* In the present study, we propose to investigate the efficacy of idiotype vaccine treatment in previously untreated patients with mantle cell lymphomas. In order to achieve minimal residual disease, patients will receive 6 cycles EPOCH chemotherapy and rituximab (EPOCH-R) followed by 5 idiotype vaccine injections.
* This study has completed accrual of 26 patients and study is closed as of 4/18/2022.

ELIGIBILITY:
* INCLUSION CRITERIA:

Tissue diagnosis of mantle cell lymphoma (confirmed in Laboratory of Pathology). Blastic cell variant will be eligible.

Age greater than or equal to 18.

Previously untreated with cytotoxic chemotherapy. Patients may have received local radiation or a short course of steroids for control of symptoms.

All stages of disease.

Lymph node of greater than or equal to 2 cm accessible for biopsy/harvest or greater than 1000/microliters of circulating tumor cells in the blood.

Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 3.

Adequate major organ function (serum creatinine 1.5 mg/dl or creatinine clearance greater than 60 ml/min; bilirubin less than 2 mg/dl (total) except less than 5 mg/dl in patients with Gilbert's syndrome as defined by greater than 80% unconjugated; absolute neutrophil count (ANC) greater than 1000 and platelets greater than 100,000) unless impairment due to organ involvement by lymphoma.

No active symptomatic ischemic heart disease, myocardial infarction or congestive heart failure within the past year. If multigated acquisition (MUGA) scan is obtained, the left ventricular ejection fraction (LVEF) should exceed 40%.

Ability to give informed consent.

EXCLUSION CRITERIA:

Antibodies to human immunodeficiency virus (HIV) or presence of hepatitis B surface antigen.

Pregnant or lactating.

Prior malignancy in past 5 years except squamous or basal cell carcinoma or curatively treated in situ of the cervix.

Involvement of central nervous system by lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-06-01 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Melani, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pittaluga S, Bijnens L, Teodorovic I, Hagenbeek A, Meerwaldt JH, Somers R, Thomas J, Noordijk EM, De Wolf-Peeters C. Clinical analysis of 670 cases in two trials of the European Organization for the Research and Treatment of Cancer Lymphoma Cooperative Group subtyped according to the Revised European-American Classification of Lymphoid Neoplasms: a comparison with the Working Formulation. Blood. 1996 May 15;87(10):4358-67. PMID 8639796
- [Background] Armitage JO. Management of mantle cell lymphoma. Oncology (Williston Park). 1998 Oct;12(10 Suppl 8):49-55. PMID 9830633
- [Background] Weisenburger DD, Armitage JO. Mantle cell lymphoma-- an entity comes of age. Blood. 1996 Jun 1;87(11):4483-94. No abstract available. PMID 8639814
- [Result] Grant C, Neelapu SS, MD2, Kwak LW, Dunleavy K, White T, Miller BW, Jaffe ES, Steinberg SM, Healey Bird B, MB, Wilson WH. Eleven-Year Follow-up of Idiotype Vaccine and DA-EPOCH-Rituximab in Untreated Mantle Cell Lymphoma: Correlation of Survival with Idiotype Immune Response. Blood (ASH Annual Meeting Abstracts) 2011 118: Abstract 2707.
- [Result] Neelapu SS, Kwak LW, Kobrin CB, Reynolds CW, Janik JE, Dunleavy K, White T, Harvey L, Pennington R, Stetler-Stevenson M, Jaffe ES, Steinberg SM, Gress R, Hakim F, Wilson WH. Vaccine-induced tumor-specific immunity despite severe B-cell depletion in mantle cell lymphoma. Nat Med. 2005 Sep;11(9):986-91. doi: 10.1038/nm1290. Epub 2005 Aug 21. PMID 16116429
- [Result] Roschewski M, Dunleavy K, Neelapu SS, Pittaluga S, Melani CJ, Jaffe ES, Shovlin M, Crossley B, Kong K, Jacob A, Kwak L, Wilson WH. Quantitative Baseline Circulating Tumor DNA Levels Correlate with GM-CSF Response to Idiotype Vaccine in Untreated Mantle Cell Lymphoma (ASH Annual Meeting Abstracts). Blood. 2016;128:2943-2943.
- [Result] Wilson WH, Neelapu S, White T, et al: Idiotype Vaccine Following EPOCH-Rituximab Treatment in Untreated Mantle Cell Lymphoma. Pro Am Soc Heme, 2002.
- [Result] Neelapu S, Wilson WH, Baskar W, et at: Induction of T-cell responses by tumor antigen vaccination in mantle cell lymphoma following rituximab-based treatment. Pro Am Soc Clin Oncol, 2003.
- [Result] Rosenwald A, Wright G, Wiestner A, Chan WC, Connors JM, Campo E, Gascoyne RD, Grogan TM, Muller-Hermelink HK, Smeland EB, Chiorazzi M, Giltnane JM, Hurt EM, Zhao H, Averett L, Henrickson S, Yang L, Powell J, Wilson WH, Jaffe ES, Simon R, Klausner RD, Montserrat E, Bosch F, Greiner TC, Weisenburger DD, Sanger WG, Dave BJ, Lynch JC, Vose J, Armitage JO, Fisher RI, Miller TP, LeBlanc M, Ott G, Kvaloy S, Holte H, Delabie J, Staudt LM. The proliferation gene expression signature is a quantitative integrator of oncogenic events that predicts survival in mantle cell lymphoma. Cancer Cell. 2003 Feb;3(2):185-97. doi: 10.1016/s1535-6108(03)00028-x. PMID 12620412
- [Result] Wilson WH, Neelapu S, Rosenwald A, et al: Idiotype Vaccine and Dose-Adjusted EPOCH-Rituximab Treatment in Untreated Mantle Cell Lymphoma: Preliminary Report on Clinical Outcome and Analysis of Immune Response. 2003, Blood 102 (11) #358.
- [Result] Fu K, Weisenburger DD, Greiner TC, Dave S, Wright G, Rosenwald A, Chiorazzi M, Iqbal J, Gesk S, Siebert R, De Jong D, Jaffe ES, Wilson WH, Delabie J, Ott G, Dave BJ, Sanger WG, Smith LM, Rimsza L, Braziel RM, Muller-Hermelink HK, Campo E, Gascoyne RD, Staudt LM, Chan WC; Lymphoma/Leukemia Molecular Profiling Project. Cyclin D1-negative mantle cell lymphoma: a clinicopathologic study based on gene expression profiling. Blood. 2005 Dec 15;106(13):4315-21. doi: 10.1182/blood-2005-04-1753. Epub 2005 Aug 25. PMID 16123218
- [Result] Wiestner A, Tehrani M, Chiorazzi M, Wright G, Gibellini F, Nakayama K, Liu H, Rosenwald A, Muller-Hermelink HK, Ott G, Chan WC, Greiner TC, Weisenburger DD, Vose J, Armitage JO, Gascoyne RD, Connors JM, Campo E, Montserrat E, Bosch F, Smeland EB, Kvaloy S, Holte H, Delabie J, Fisher RI, Grogan TM, Miller TP, Wilson WH, Jaffe ES, Staudt LM. Point mutations and genomic deletions in CCND1 create stable truncated cyclin D1 mRNAs that are associated with increased proliferation rate and shorter survival. Blood. 2007 Jun 1;109(11):4599-606. doi: 10.1182/blood-2006-08-039859. Epub 2007 Feb 13. PMID 17299095
- [Result] Dunleavy K, Neelapu SS, Kwak LW, Grant C, Santos CF, Popa M, White T, Miller B, Jaffe ES, Steinberg SM and Wilson WH. Association of idiotype vaccine-induced T-cell response with improved survival and time-to-next treatment (TTNT) in untreated mantle cell lymphoma (MCL). Journal of Clinical Oncology, 2012 ASCO Annual Meeting Proceedings (Post-Meeting Edition).Vol 30, No 15_suppl (May 20 Supplement), 2012: 2528.
- [Derived] Lai C, Cole DE, Steinberg SM, Lucas N, Dombi E, Melani C, Roschewski M, Balis F, Widemann BC, Wilson WH. Doxorubicin pharmacokinetics and toxicity in patients with aggressive lymphoma and hepatic impairment. Blood Adv. 2023 Feb 28;7(4):529-532. doi: 10.1182/bloodadvances.2022007431. PMID 35882475
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-C-0133.html

RESULTS

PARTICIPANT FLOW:
Period: EPOCH-R Administration
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Started | 26
Completed | 26 (26 completed the EPOCH-R treatment and 23/26 moved on to vaccine treatment.)
Not Completed | 0
Period: Vaccine Administration Following EPOCH-R
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Started | 24
Completed | 23
Not Completed | 1
Not completed — Participant progressed before receiving the last vaccine. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 57 [22 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
Mantle Cell Lymphoma International Prognostic Index (MIPI) [Count of Participants; unit: Participants] — MIPI is a prognostic score (i.e., risk groups) for participants with mantle cell lymphoma. Low- risk scores (i.e., 0-3) indicate better survival and high-risk scores (i.e., 6-11) indicate lower survival. Intermediate-risk scores (i.e., 4-5) is neither low nor high with intermediate survival.
  Participants
    Low | 16
    Intermediate | 7
    High | 3
Performance Status [Median (Full Range); unit: score on a scale] — ECOG score is an indication of a participant's functional status. An ECOG score of 0 indicates a participant is fully active without any performance restrictions. An ECOG score of 1 indicates a participant is restricted in physically strenuous activity but ambulatory and able to carry out light work. An ECOG score of 2 indicates a participant is capable of self-care but unable to carry out any work activities and is up and about greater than 50% of waking hours.
  score on a scale | 1 [0 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS) in Participants Treated With Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (EPOCH-R)
Description: PFS is time from on study date until disease relapse or progression, death, or date of last follow-up. Progression was measured by the International Workshop to Standardize Response Criteria for non-Hodgkin's Lymphoma and is defined as ≥50% increase from nadir in the sum of the products of the greatest diameters (SPD) of any previously involved node or the appearance of any new lesion.
Time Frame: From participants on study date until date of disease relapse or progression, death, or date of last follow-up, assessed up to 245.8 months
Measure: Median (Full Range); unit: Months
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 26
Months | 23.5 [8.8 to 245.8]

2. Primary Outcome: Percentage of Participants With an Antibody Response to Idiotype Vaccine
Description: Participants with an immune response to idiotype vaccine measured by enzyme-linked immunosorbent assay (ELISA) to detect antibody binding to tumor cells. Positive response was defined as at least a fourfold increase in antibody titer.
Time Frame: Weeks 12 to 32
Population: 23/26 participants were analyzed because vaccine was unable to be produced in two participants and one participant progressed prior to receiving the last vaccine dose.
Measure: Number; unit: percentage of participants
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 23
percentage of participants | 30

3. Secondary Outcome: Percentage of Participants Whose Cancer Shrinks or Disappears After Treatment With Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (EPOCH-R)
Description: Response was measured by the International Workshop to Standardize Response Criteria for non-Hodgkin's Lymphoma. Complete Response (CR) is a complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities (e.g., Lactate dehydrogenase (LDH) definitely assignable to the lymphoma. Complete Response Unconfirmed (CRu) is as per CR criteria except that if a residual node is > 1.5cm, it must have regressed by > 75% in the sum of the products of the greatest diameters (SPD). Partial Response (PR) is ≥50% decreased in the SPD of 6 largest dominant nodes or nodal masses. Stable Disease (SD) is defined as less than a PR but not progressive disease. Progression is ≥50% increase from nadir in the SPD of any previously involved node or the appearance of any new lesion.
Time Frame: After 6 cycles of EPOCH-R therapy, an average of 18 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 26
percentage of participants
  Complete Response | 80.8
  Complete Response Unconfirmed | 7.7
  Partial Response | 7.7
  Stable Disease | 0
  Progression | 3.8

4. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Serious and/or Non-serious Toxicity That Occurred That is at Least Possibly Related to Drug or Vaccine
Description: Serious and/or non-serious adverse events were assessed by the Common Toxicity Criteria (CTC v2.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: Up to 30 days after last intervention, up to 12.5 months or 1.04 years
Measure: Number; unit: percentage of participants
Groups:
- Grade 3: Grade 3 is severe.
- Grade 4: Grade 4 is life-threatening.
- Grade 5: Grade 5 is death related to adverse event.
Arm/Group | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 26 | 26 | 26
percentage of participants
  Allergic reaction | 3.8 | 0 | 0
  Anemia | 69.2 | 3.8 | 0
  Febrile neutropenia | 42.3 | 3.8 | 0
  Leukopenia | 0 | 84.6 | 0
  Lymphopenia | 38.5 | 0 | 0
  Neutropenia | 0 | 88.5 | 0
  Thrombocytopenia | 50 | 7.7 | 0
  Thrombosis | 15.4 | 0 | 0
  Infusion related reaction | 3.8 | 0 | 0
  Serum glutamic oxaloacetic transaminase (SGOT) elevation | 3.8 | 0 | 0
  Serum glutamic pyruvic transaminase (SGPT) elevation | 3.8 | 0 | 0
  Infection | 15.4 | 3.8 | 0
  Hyperglycemia | 3.8 | 0 | 0
  Hypomagnesemia | 3.8 | 0 | 0
  Cerebrovascular ischemia | 0 | 3.8 | 0
  Motor neuropathy | 11.5 | 0 | 0
  Sensory neuropathy | 3.8 | 0 | 0
  Back pain | 3.8 | 0 | 0
  Dyspnea | 3.8 | 0 | 0
  Erectile dysfunction | 3.8 | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS was determined by the Kaplan-Meier method and is defined as the time from treatment start date until date of death or last follow-up.
Time Frame: Time from treatment start date until date of death or date last follow-up, up to 250 months
Measure: Median (Full Range); unit: Months
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 26
Months | 89.7 [32.4 to 245.8]

6. Secondary Outcome: Progression Free Survival (PFS) in Participants Who Received Idiotype Vaccine
Description: PFS is defined as the time from start of treatment until disease relapse or progression, death, or last follow-up. Progression was measured by the International Workshop to Standardize Response Criteria for non-Hodgkin's Lymphoma and is defined as ≥50% increase from nadir in the sum of the products of the greatest diameters (SPD) of any previously involved node or the appearance of any new lesion
Time Frame: Time from treatment start date until date of disease relapse or progression, death, or date last follow-up, an average of 25 months
Population: 23/26 participants were analyzed because vaccine was unable to be produced in two participants and one participant progressed prior to receiving the last vaccine.
Measure: Median (Full Range); unit: Months
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 23
Months | 25.0 [8.8 to 245.8]

7. Secondary Outcome: Percentage of Participants With Antibodies to Keyhole Limpet Haemocyanin (KLH)
Description: Participants with an immune response against carrier molecule KLH measured by enzyme-linked immunosorbent assay (ELISA) to detect antibody binding to tumor cells. Positive response was defined as at least a fourfold increase in antibody titer.
Time Frame: After vaccinations administered at 0, 1, 2, 3 and 5 months
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 23
percentage of participants | 74

8. Secondary Outcome: Percentage of Participants With Induction of Type 1 Cytokine T-cell Response
Description: Participants with tumor specific T-cell responses during B-cell recovery was assessed in a Clinical Laboratory Improvement Amendments (CLIA) certified lab and were measured by flow cytometry and/or enzyme-linked immunosorbent spot (ELISPOT). A positive response required the response to be at least twice the negative controls.
Time Frame: After vaccinations administered at 0, 1, 2, 3 and 5 months
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 23
percentage of participants
  Peripheral blood mononuclear cells (PBMC) | 87
  Granulocyte macrophage colony-stimulating factor (GM-CSF) | 65
  Tumor necrosis factor α (TNFα) | 52
  Interferon-gamma (IFN-γ) | 74

9. Secondary Outcome: Time to Recovery of CD4 T Lymphocytes (CD4+)
Description: Recovery of CD4+ was measured by flow cytometry. Blood samples were collected via apheresis and analyzed by multicolor flow cytometry in peripheral blood mononuclear cells (PBMCs) for cluster of differentiation 4 (CD4). Time to recovery of CD4 T lymphocytes was defined as the time required for CD4 T lymphocytes to increase above the lower limit of normal of the normal laboratory value range of 359 cells/mcL
Time Frame: After chemotherapy before vaccination, up to 6 months
Measure: Median (Full Range); unit: Months
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 23
Months | 3 [2.8 to 5.4]

10. Other Pre Specified Outcome: Here is the Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Toxicity Criteria (CTC v2.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Toxicity Criteria (CTC v2.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Up to 30 days after last intervention, up to 12.5 months or 1.04 years
Measure: Count of Participants; unit: Participants
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
Number analyzed (Participants) | 26
Participants | 26

ADVERSE EVENTS:
Time Frame: Up to 30 days after last intervention, up to 12.5 months or 1.04 years for serious and/or non-serious adverse events and up to 250 months for all-cause mortality.
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab
All-Cause Mortality (participants affected / at risk) | 17/26
Serious Adverse Events (participants affected / at risk) | 14/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (N=26)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 10 (10)
Infection (Infections and infestations) | 2 (2)
Infusion related reaction (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (N=26)
Death unrelated to research and related to disease progression (General disorders) | 17 (17)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Alkaline phosphatase elevation (Hepatobiliary disorders) | 7 (7)
Allergic reaction (Immune system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (21)
Anemia (Blood and lymphatic system disorders) | 24 (24)
Anorexia (Gastrointestinal disorders) | 14 (14)
Anxiety (Psychiatric disorders) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bilirubin elevation (Hepatobiliary disorders) | 1 (1)
Blurred vision (Eye disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 23 (23)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Cerebrovascular ischemia (Cardiac disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 25 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12)
CPK elevation (Metabolism and nutrition disorders) | 1 (1)
Creatinine elevation (Renal and urinary disorders) | 1 (1)
Decreased libido (Reproductive system and breast disorders) | 1 (1)
Depression (Nervous system disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 19 (19)
Dizziness (Nervous system disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dysuria (Renal and urinary disorders) | 2 (2)
Edema (Cardiac disorders) | 7 (7)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Euphoria (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 25 (25)
Febrile neutropenia (Infections and infestations) | 12 (12)
Fever (General disorders) | 5 (5)
Floaters (Eye disorders) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Gynecomastia (Endocrine disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (10)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hot flashes (Endocrine disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hypothyroid (Endocrine disorders) | 1 (1)
Infection (Infections and infestations) | 6 (6)
Infusion related reaction (General disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Leg pain (General disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 22 (22)
Lymphopenia (Blood and lymphatic system disorders) | 13 (13)
Motor neuropathy (Nervous system disorders) | 5 (5)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 10 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14)
Nausea (Gastrointestinal disorders) | 14 (14)
Neutropenia (Blood and lymphatic system disorders) | 23 (23)
Phlebitis (Cardiac disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
PT elevation (Blood and lymphatic system disorders) | 1 (1)
PTT elevation (Blood and lymphatic system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Sensory neuropathy (Nervous system disorders) | 25 (25)
SGOT elevation (Hepatobiliary disorders) | 5 (5)
SGPT elevation (Hepatobiliary disorders) | 5 (5)
Stomatitis (Gastrointestinal disorders) | 24 (24)
Taste disturbance (Gastrointestinal disorders) | 17 (17)
Tearing (Eye disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (22)
Thrombosis (Cardiac disorders) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1)
Visual loss (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7)
Weight loss (General disorders) | 6 (6)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT00005780/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT00005780/ICF_001.pdf